CLINICAL TRIAL: NCT02473159
Title: Clinical Application of Near-infrared Fluorescence Guided Localization on Breast Surgery in Breast Cancer: Interventional Pilot Study for 5 Patients
Brief Title: Clinical Application of Near-infrared Fluorescence Guided Localization on Breast Surgery in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, So-Youn Jung, Medical Doctor, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-1410202-2
Record Dates: First submitted 2015-05-08; First posted 2015-06-16 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Near-infrared fluorescence; Indocyanine green, ICG; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- indocyanine green (Experimental): As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
  Other Names: Near-infrared fluorescence

SUMMARY:
Near-infrared (NIR) fluorescence imaging using indocyanine green (ICG) has been used for breast cancer surgery such as sentinel lymph node (SLN) mapping and breast cancer localization.

In this study, our hypothesis are as following:

1. As inject only indocyanine green (ICG), it provide the surgeon visual guidance to ensure better outcome.
2. indocyanine green (ICG) permitted accurate preoperative and intraoperative detection of the SLNs as well as nonpalpable benign brest lesion in patients with breast cancer.

DETAILED DESCRIPTION:
Indocyanine green, ICG (ICG-fluorescence)

* ICG is the most commonly used fluorophore which approve by FDA.
* NIR-F imaging with ICG could be used in various surgeries. For example, SLN mapping in breast cancer and localization of liver metastasis, especially superficial lesion
* Contains sodium iodide, patients who have history of allergy to iodides should be used as caution.

Nonpalpable benign brest lesion localization

* New method for the localization and resection of non-palpable breast lesions.
* The breast lesion was correctly localized, and the area of ICG corresponded well to the site of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* nonpalpable breast tumor ≤ 2cm in patients with breast cancer.
* patients who need breast biopsy as treatment for breast cancer.
* Eastern Cooperative Oncology Group Performance status 0 or 1
* consented patients with more than 20 years, less than 70 years

Exclusion Criteria:

* nonpalpable breast tumor ≥ 2cm in patients with breast cancer.
* pregnancy
* history of severe allergy to ICG(Indocyanine Green)
* iode hypersensitiveness

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
detection rate | one day
  after complete resection with intraoperative ultrasound confirmed the lesion

SECONDARY OUTCOMES:
determine the pathological stability | one day
  determine the pathological stability with biopsy results confirmed during surgery

OTHER OUTCOMES:
detection rate and reoperation rate | participants will be followed for the duration of return to clinic, an expected average of 1 weeks
  tumor detection rate and reoperation rate of resection margin

CONTACTS AND LOCATIONS:
Overall Officials: So-Youn Jung, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea